CLINICAL TRIAL: NCT07064746
Title: Clinical Application Study of [123I]Metaiodobenzylguanidine and Somatostatin Receptor-Targeted Imaging in the Diagnosis and Staging of Neuroblastoma
Acronym: MIBG & SSTR NB
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Jiangsu Province Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY20220701-01
Record Dates: First submitted 2025-07-06; First posted 2025-07-15 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma (NB)
Keywords: neuroblastoma; SSTR; MIBG; PET
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Neuroblastoma Imaging Cohort: This cohort includes pediatric patients (≤18 years) with suspected or confirmed neuroblastoma. Interventions include diagnostic imaging with ¹²³I-MIBG SPECT/CT and SSTR PET/CT for staging, therapy planning, and disease monitoring.
  Interventions: Diagnostic Test: ¹²³I-MIBG SPECT/CT; Diagnostic Test: SSTR PET

INTERVENTIONS:
Diagnostic Test: ¹²³I-MIBG SPECT/CT — Patients take Lugol's iodine 2 days and on the day of injection for thyroid blockade. ¹²³I-MIBG (3-5 MBq/kg; max 370 MBq) is given IV. Whole-body planar imaging is performed 24 h post-injection, then focused SPECT/CT of any suspicious areas with low-dose CT; children are sedated only if motion control is required.
Diagnostic Test: SSTR PET — Patients receive an intravenous bolus of 68Ga-DOTA-TATE (1.8-2.2 MBq/kg, max 200 MBq). After a 45-60 min uptake phase, a low-dose whole-body PET/CT or PET/MRI (skull base-mid-thigh) is acquired for ~20 min; MRI or CT provides attenuation correction. Sedation used when required.

SUMMARY:
The goal of this prospective observational study is to evaluate the diagnostic performance of ¹²³I-MIBG SPECT/CT and SSTR PET in Chinese children with suspected or confirmed neuroblastoma (NB). The main questions it aims to answer are:

* What are the sensitivity and specificity of each modality-alone and combined-for initial staging and for detecting relapse or metastasis?
* Can SSTR-targeted PET reliably identify MIBG-negative NB lesions and help select candidates for peptide-receptor radionuclide therapy (PRRT)?

Pediatric patients (≤18 years) undergoing routine evaluation for NB will receive both imaging studies; results will be correlated with histopathology, clinical course, and 24-month follow-up.

DETAILED DESCRIPTION:
Neuroblastoma (NB) is the most common extracranial solid tumor in children. More than 50 % of cases occur before the age of two, while diagnoses after 10 years old are rare. NB accounts for approximately 6 - 10 % of pediatric malignancies. Its biological behavior is highly heterogeneous, with diverse molecular features, a high risk of metastasis, and often occult primary sites, making early detection and definitive diagnosis difficult [1-3]. Rapid disease progression further complicates treatment.

In recent years, driven by large international multicenter collaborations, the diagnosis and management of pediatric NB have entered an era of molecular imaging and targeted theranostics. Especially overseas, rapid advances in screening, diagnosis, treatment research, and clinical translation have yielded well-established guidelines and consensus statements, markedly improving the 5-year survival rate [4]. In contrast, research and clinical translation in China lag behind, and understanding of NB biology varies across regions, leading to uneven diagnostic and therapeutic levels without unified protocols. As a result, an increasing number of Chinese patients seek molecular imaging and targeted therapy abroad. Accelerating domestic translation of new NB technologies is thus critical to improving outcomes.

Nuclear medicine imaging (molecular imaging) employs radionuclide-labeled tracers for early lesion detection. For NB, modalities include classic radioiodinated metaiodobenzylguanidine (MIBG) imaging (¹³¹I/¹²³I/¹²⁴I-MIBG, ¹⁸F-MFBG), ¹⁸F-FDG metabolic imaging, somatostatin-receptor (SSTR)-targeted imaging (⁶⁸Ga-DOTA-TATE/TOC/NOC peptides), and ¹⁸F-DOPA imaging. With continual upgrades of SPECT/CT, quantitative SPECT/CT, and PET/CT-MRI, comparative studies on diagnostic accuracy, staging, early detection of relapse/metastasis, radiation safety, and therapy response assessment have flourished. International indications for NB radionuclide imaging include [5-7]: confirmation of suspected NB/pheochromocytoma/ganglioneuroma, disease staging, treatment planning and response evaluation, post-therapy follow-up, and selection for radionuclide therapy.

NB cells overexpress the norepinephrine transporter; hence norepinephrine analogs such as MIBG are ideal imaging (and therapeutic) ligands. Radioiodinated MIBG accumulates in neural-crest-derived tissues and tumors, exhibiting high sensitivity (88-92 %) and specificity (83-92 %) [8]. It distinguishes residual tumor from non-specific findings on anatomic imaging and more accurately evaluates bone marrow metastases than MRI [10, 11]. ¹³¹I-MIBG is widely used therapeutically, and post-therapy ¹³¹I-MIBG scans assess tracer uptake, disease status, and predict response, forming part of theranostic guidelines [8, 9, 12-14]. However, ¹³¹I emits high-energy γ-photons (364 keV) and has a long half-life, resulting in poorer SPECT image quality and lower sensitivity than ¹²³I (159 keV, much shorter half-life). The shorter half-life of ¹²³I permits higher administered activity within the same radiation dose, yielding superior images [15]. Consequently, ¹²³I-MIBG is expected to become the optimal screening tool for selecting patients for ¹³¹I-MIBG therapy. In high-risk NB, ¹²³I-MIBG detects recurrent bone metastases in 94 % of cases versus 43 % for ¹⁸F-FDG PET/CT [9, 10]. MIBG imaging remains the standard for staging and treatment assessment [16-18].

About 10 % of NBs show low or absent MIBG uptake, risking false-negative results. Combining modalities helps overcome this limitation. Somatostatin, a hypothalamic peptide that inhibits pituitary growth hormone and gastrointestinal hormones [19-21], binds receptors found on pancreatic, neuroendocrine, meningeal, and breast tumors [21-24]. High-affinity SSTRs are expressed in 77-89 % of NB cells [25-28]. Numerous ⁶⁸Ga-DOTA peptides target SSTRs, such as ⁶⁸Ga-DOTA-TATE (highest affinity for SSTR2), ⁶⁸Ga-DOTA-TOC (SSTR5), and ⁶⁸Ga-DOTA-NOC (SSTR3 and SSTR5) [29]. Compared with ¹²³/¹³¹I-MIBG, SSTR-PET/CT offers advantages: faster plasma clearance (2 h vs 2 days), same-day injection and imaging, shorter ⁶⁸Ga half-life (68 min vs 13.1 h/8 days), rapid acquisition (20-40 min vs ~1 h), and minimal preparation (no Lugol's solution). One study showed ⁶⁸Ga-DOTA-TOC PET/CT sensitivity of 94.4 %, significantly higher than ¹²³I-MIBG (76.9 %).

Systematic data on MIBG and SSTR imaging in Chinese NB are scarce. Peptide receptor radionuclide therapy (PRRT) with agents like ¹⁷⁷Lu-DOTA-TATE-proven feasible and safe abroad [30, 31]-is attractive, offering outpatient treatment without thyroid blockade, simplifying care for children and families. Small studies have applied PRRT to relapsed pediatric NB [32-35].

Given tumor heterogeneity, different molecular probes deliver complementary diagnostic and therapeutic information. Although combination imaging is well studied internationally, domestic data are lacking. Ethnic and regional factors warrant investigation. This study will employ ¹²³I-MIBG SPECT/CT fusion and SSTR PET/CT or(and) MRI for NB diagnosis, staging, and follow-up, aiming to provide valuable insights for early definitive diagnosis, precise staging, radionuclide-targeted therapy, and response evaluation in Chinese patients. In heterogeneous tumors, multimodal imaging is expected to offer clear advantages for staging, phenotype characterization, prognostication, and treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 0-18 years, any sex
2. Histologically confirmed or clinically highly suspected neuroblastoma with planned imaging assessment
3. At least one measurable lesion on conventional imaging such as CT or MRI
4. ECOG performance status 0-2 and an expected survival of ≥3 months
5. Hematologic, hepatic, and renal function meeting the following criteria: Hb ≥ 90 g/L, ANC ≥ 1.5 × 10⁹/L, platelets ≥ 100 × 10⁹/L, ALT/AST ≤ 2.5 × ULN, Cr ≤ 1.5 × ULN
6. Informed consent signed by the subject or legal guardian

Exclusion Criteria:

1. Known history of severe allergy to the radioactive isotope or molecular probe components to be used;
2. Pregnancy or lactation;
3. Receipt of high-dose chemotherapy/radiotherapy, radionuclide therapy, or participation in other interventional clinical trials within the past 4 weeks;
4. Severe or uncontrolled cardiac, pulmonary, hepatic, or renal insufficiency, or active severe infection;
5. Bone marrow suppression not yet recovered (Hb < 90 g/L, ANC < 1.5 × 10⁹/L, platelets < 100 × 10⁹/L);
6. Inability to complete imaging examinations such as PET/CT (e.g., severe claustrophobia, inability to lie supine for ≥ 30 min);
7. Any other situation deemed inappropriate for enrollment by the investigator.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Target population
  * Consecutively enrolled neuroblastoma (NB) patients aged 0-18 years, of any sex;
  * Inclusive of all INSS stages Ⅰ-ⅣS and risk groups (low, intermediate, high), covering newly diagnosed, relapsed, and refractory cases;
  * Pathologically confirmed NB, or highly suspected NB based on characteristic imaging plus elevated urinary VMA/HVA, with at least one measurable lesion on routine CT/MRI;
  * Primary and metastatic cases (bone, bone marrow, liver, lymph nodes, etc.) at different treatment stages (before treatment, during treatment, follow-up) are allowed to ensure representativeness in age, sex, histology, stage, and metastatic site distribution.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
SUVmean | baseline and 6 months
  SUVmean is obtained by outlining a 3-D volume-of-interest around the lesion on attenuation-corrected PET images and averaging all voxel values. Standardized uptake values are calculated as voxel activity concentration (kBq/mL) divided by injected activity per body weight (kBq/g).
SUVmax | Baseline and 6 months
  SUVmax is obtained by outlining a 3-D volume of interest (VOI) around the lesion on attenuation-corrected PET images; the software reports the single voxel with the highest activity concentration, normalized to injected tracer dose divided by the patient's body weight (MBq/kg).
SUVpeak | baseline and 6 months
  SUVpeak is obtained by drawing a fixed-size, 1 cm³ spherical volume of interest centered on the hottest voxel within the tumor on attenuation-corrected PET images; the mean activity concentration inside this sphere is normalized to injected dose per body weight to yield SUVpeak, minimizing noise while reflecting maximal metabolic activity.

CONTACTS AND LOCATIONS:
Overall Officials: Guoqiang Shao, Dr, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Within 6 months of the end of the trial, trial data are uploaded to http://www.medresman.org.cn/login.aspx
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 6 months and ending 3 years after the publication of results
Access Criteria: Qualified academic investigators with an IRB-approved proposal may request access to de-identified individual participant data (IPD), the full study protocol, blank case report forms, and the English/Chinese informed-consent templates. Requests should be emailed to the corresponding author; after signing a data-sharing agreement, files will be shared through a secure, password-protected institutional repository within 30 days.
URL: http://www.medresman.org.cn/login.aspx

REFERENCES:
- [Background] Menda Y, O'Dorisio MS, Kao S, Khanna G, Michael S, Connolly M, Babich J, O'Dorisio T, Bushnell D, Madsen M. Phase I trial of 90Y-DOTATOC therapy in children and young adults with refractory solid tumors that express somatostatin receptors. J Nucl Med. 2010 Oct;51(10):1524-31. doi: 10.2967/jnumed.110.075226. Epub 2010 Sep 16. PMID 20847174
- [Background] Sadowski SM, Neychev V, Millo C, Shih J, Nilubol N, Herscovitch P, Pacak K, Marx SJ, Kebebew E. Prospective Study of 68Ga-DOTATATE Positron Emission Tomography/Computed Tomography for Detecting Gastro-Entero-Pancreatic Neuroendocrine Tumors and Unknown Primary Sites. J Clin Oncol. 2016 Feb 20;34(6):588-96. doi: 10.1200/JCO.2015.64.0987. Epub 2015 Dec 28. PMID 26712231
- [Background] Gains JE, Bomanji JB, Fersht NL, Sullivan T, D'Souza D, Sullivan KP, Aldridge M, Waddington W, Gaze MN. 177Lu-DOTATATE molecular radiotherapy for childhood neuroblastoma. J Nucl Med. 2011 Jul;52(7):1041-7. doi: 10.2967/jnumed.110.085100. Epub 2011 Jun 16. PMID 21680680
- [Background] Kong G, Hofman MS, Murray WK, Wilson S, Wood P, Downie P, Super L, Hogg A, Eu P, Hicks RJ. Initial Experience With Gallium-68 DOTA-Octreotate PET/CT and Peptide Receptor Radionuclide Therapy for Pediatric Patients With Refractory Metastatic Neuroblastoma. J Pediatr Hematol Oncol. 2016 Mar;38(2):87-96. doi: 10.1097/MPH.0000000000000411. PMID 26296147
- [Background] Hofman MS, Lau WF, Hicks RJ. Somatostatin receptor imaging with 68Ga DOTATATE PET/CT: clinical utility, normal patterns, pearls, and pitfalls in interpretation. Radiographics. 2015 Mar-Apr;35(2):500-16. doi: 10.1148/rg.352140164. PMID 25763733
- [Background] Georgantzi K, Tsolakis AV, Stridsberg M, Jakobson A, Christofferson R, Janson ET. Differentiated expression of somatostatin receptor subtypes in experimental models and clinical neuroblastoma. Pediatr Blood Cancer. 2011 Apr;56(4):584-9. doi: 10.1002/pbc.22913. Epub 2010 Nov 30. PMID 21298743
- [Background] Moertel CL, Reubi JC, Scheithauer BS, Schaid DJ, Kvols LK. Expression of somatostatin receptors in childhood neuroblastoma. Am J Clin Pathol. 1994 Dec;102(6):752-6. doi: 10.1093/ajcp/102.6.752. PMID 7801887
- [Background] Albers AR, O'Dorisio MS, Balster DA, Caprara M, Gosh P, Chen F, Hoeger C, Rivier J, Wenger GD, O'Dorisio TM, Qualman SJ. Somatostatin receptor gene expression in neuroblastoma. Regul Pept. 2000 Mar 17;88(1-3):61-73. doi: 10.1016/s0167-0115(99)00121-4. PMID 10706954
- [Background] O'Dorisio MS, Chen F, O'Dorisio TM, Wray D, Qualman SJ. Characterization of somatostatin receptors on human neuroblastoma tumors. Cell Growth Differ. 1994 Jan;5(1):1-8. PMID 8123588
- [Background] Orlando C, Raggi CC, Bianchi S, Distante V, Simi L, Vezzosi V, Gelmini S, Pinzani P, Smith MC, Buonamano A, Lazzeri E, Pazzagli M, Cataliotti L, Maggi M, Serio M. Measurement of somatostatin receptor subtype 2 mRNA in breast cancer and corresponding normal tissue. Endocr Relat Cancer. 2004 Jun;11(2):323-32. doi: 10.1677/erc.0.0110323. PMID 15163307
- [Background] Reubi JC, Maurer R, Klijn JG, Stefanko SZ, Foekens JA, Blaauw G, Blankenstein MA, Lamberts SW. High incidence of somatostatin receptors in human meningiomas: biochemical characterization. J Clin Endocrinol Metab. 1986 Aug;63(2):433-8. doi: 10.1210/jcem-63-2-433. PMID 3013920
- [Background] Reubi JC, Maurer R, von Werder K, Torhorst J, Klijn JG, Lamberts SW. Somatostatin receptors in human endocrine tumors. Cancer Res. 1987 Jan 15;47(2):551-8. PMID 3024822
- [Background] Lamberts SW, Koper JW, Reubi JC. Potential role of somatostatin analogues in the treatment of cancer. Eur J Clin Invest. 1987 Aug;17(4):281-7. doi: 10.1111/j.1365-2362.1987.tb02188.x. No abstract available. PMID 2889601
- [Background] Reichlin S. Somatostatin. N Engl J Med. 1983 Dec 15;309(24):1495-501. doi: 10.1056/NEJM198312153092406. No abstract available. PMID 6139753
- [Background] Burgus R, Ling N, Butcher M, Guillemin R. Primary structure of somatostatin, a hypothalamic peptide that inhibits the secretion of pituitary growth hormone. Proc Natl Acad Sci U S A. 1973 Mar;70(3):684-8. doi: 10.1073/pnas.70.3.684. PMID 4514982
- [Background] Matthay KK, Shulkin B, Ladenstein R, Michon J, Giammarile F, Lewington V, Pearson AD, Cohn SL. Criteria for evaluation of disease extent by (123)I-metaiodobenzylguanidine scans in neuroblastoma: a report for the International Neuroblastoma Risk Group (INRG) Task Force. Br J Cancer. 2010 Apr 27;102(9):1319-26. doi: 10.1038/sj.bjc.6605621. PMID 20424613
- [Background] Leung A, Shapiro B, Hattner R, Kim E, de Kraker J, Ghazzar N, Hartmann O, Hoefnagel CA, Jamadar DA, Kloos R, Lizotte P, Lumbroso J, Rufini V, Shulkin BL, Sisson JC, Thein A, Troncone L. Specificity of radioiodinated MIBG for neural crest tumors in childhood. J Nucl Med. 1997 Sep;38(9):1352-7. PMID 9293786
- [Background] Vik TA, Pfluger T, Kadota R, Castel V, Tulchinsky M, Farto JC, Heiba S, Serafini A, Tumeh S, Khutoryansky N, Jacobson AF. (123)I-mIBG scintigraphy in patients with known or suspected neuroblastoma: Results from a prospective multicenter trial. Pediatr Blood Cancer. 2009 Jul;52(7):784-90. doi: 10.1002/pbc.21932. PMID 19185008
- [Background] Liu B, Zhuang H, Servaes S. Comparison of [123I]MIBG and [131I]MIBG for imaging of neuroblastoma and other neural crest tumors. Q J Nucl Med Mol Imaging. 2013 Mar;57(1):21-8. PMID 23474632
- [Background] Olivier P, Colarinha P, Fettich J, Fischer S, Frokier J, Giammarile F, Gordon I, Hahn K, Kabasakal L, Mann M, Mitjavila M, Piepsz A, Porn U, Sixt R, van Velzen J. Guidelines for radioiodinated MIBG scintigraphy in children. Eur J Nucl Med Mol Imaging. 2003 May;30(5):B45-50. doi: 10.1007/s00259-003-1138-9. Epub 2003 Mar 26. PMID 12658506
- [Background] Bombardieri E, Giammarile F, Aktolun C, Baum RP, Bischof Delaloye A, Maffioli L, Moncayo R, Mortelmans L, Pepe G, Reske SN, Castellani MR, Chiti A; European Association for Nuclear Medicine. 131I/123I-metaiodobenzylguanidine (mIBG) scintigraphy: procedure guidelines for tumour imaging. Eur J Nucl Med Mol Imaging. 2010 Dec;37(12):2436-46. doi: 10.1007/s00259-010-1545-7. PMID 20644928
- [Background] Ohdaira H, Sasaki T, Yoshida K. A subset of microRNAs potentially acts as a convergent hub for upstream transcription factors in cancer cells. Oncol Rep. 2010 Nov;24(5):1371-81. doi: 10.3892/or_00000995. PMID 20878133
- [Background] Frazier AA. Radiologic-Pathologic Features to Discern Nonepithelial versus Epithelial Pancreatic Tumors. Radiographics. 2016 Jan-Feb;36(1):122. doi: 10.1148/rg.2016154023. No abstract available. PMID 26761534
- [Background] Sharp SE, Shulkin BL, Gelfand MJ, Salisbury S, Furman WL. 123I-MIBG scintigraphy and 18F-FDG PET in neuroblastoma. J Nucl Med. 2009 Aug;50(8):1237-43. doi: 10.2967/jnumed.108.060467. Epub 2009 Jul 17. PMID 19617326
- [Background] Taggart DR, Han MM, Quach A, Groshen S, Ye W, Villablanca JG, Jackson HA, Mari Aparici C, Carlson D, Maris J, Hawkins R, Matthay KK. Comparison of iodine-123 metaiodobenzylguanidine (MIBG) scan and [18F]fluorodeoxyglucose positron emission tomography to evaluate response after iodine-131 MIBG therapy for relapsed neuroblastoma. J Clin Oncol. 2009 Nov 10;27(32):5343-9. doi: 10.1200/JCO.2008.20.5732. Epub 2009 Oct 5. PMID 19805691
- [Background] Giammarile F, Chiti A, Lassmann M, Brans B, Flux G; EANM. EANM procedure guidelines for 131I-meta-iodobenzylguanidine (131I-mIBG) therapy. Eur J Nucl Med Mol Imaging. 2008 May;35(5):1039-47. doi: 10.1007/s00259-008-0715-3. PMID 18274745
- [Background] Shulkin BL, Shapiro B. Current concepts on the diagnostic use of MIBG in children. J Nucl Med. 1998 Apr;39(4):679-88. PMID 9544682
- [Background] Sharp SE, Trout AT, Weiss BD, Gelfand MJ. MIBG in Neuroblastoma Diagnostic Imaging and Therapy. Radiographics. 2016 Jan-Feb;36(1):258-78. doi: 10.1148/rg.2016150099. PMID 26761540